CLINICAL TRIAL: NCT01204086
Title: Pharmacogenomics Studies of Antidepressants
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: Department of Health, Executive Yuan, R.O.C. (Taiwan) (Other Government)
Responsible Party: Po See Chen/ MD, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HR-95-06; DOH96-TD-D-113-041 (Other Grant/Funding Number: Department of Health, Taiwan)
Record Dates: First submitted 2010-09-15; First posted 2010-09-17 (Estimated); Last update posted 2010-09-17 (Estimated); Status verified 2010-09

CONDITIONS: Major Depressive Disorder; Antidepressive Agents; Pharmacogenetics; Venlafaxine; Fluoxetine
Keywords: Major Depressive Disorder; Antidepressants; Pharmacogenetics; venlafaxine; fluoxetine
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Venlafaxine Hydrochloride; Fluoxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- venlafaxine (Experimental)
  Interventions: Drug: Venlafaxine
- fluoxetine (Experimental)
  Interventions: Drug: Fluoxetine

INTERVENTIONS:
Drug: Venlafaxine — The initial dose of venlafaxine was 37.5 mg once daily for 4 days titrated to 75 mg once daily, which could be increased by 75 mg in divided doses to a maximal daily dose of 225 mg.
  Arms: venlafaxine
Drug: Fluoxetine — The initial dose of fluoxetine was 20 mg once daily, which could be increased by 20 mg in divided doses to a maximal daily dose of 80 mg.
  Arms: fluoxetine

SUMMARY:
The purpose of this study is to establish the clinical effectiveness of antidepressants by pharmacogenomic approach, and to determine the levels of inflammatory factors between the baseline and the end point of the study in Taiwanese major depressive disorder (MDD) patients.

ELIGIBILITY:
Inclusion Criteria:

* Age: 16-65 years old
* Signed informed consent by patient or legal representative
* Hamilton Rating Scale for Depression (HDRS) scores ≥ 16
* A diagnosis of MDD according to DSM-IV criteria made by a specialist in psychiatry

Exclusion Criteria:

* monoamine oxidase inhibitor or antidepressant treatment within two weeks prior to entering the study
* A DSM-IV diagnosis of substance abuse within the past three months
* An organic mental disease, mental retardation or dementia
* A serious surgical condition or physical illness
* Patients who were pregnant or breastfeeding

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-03; Primary Completion 2010-12 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale (HDRS) | baseline
Hamilton Depression Rating Scale (HDRS) | 2 weeks
Hamilton Depression Rating Scale (HDRS) | 4 weeks
Hamilton Depression Rating Scale (HDRS) | 6 weeks

SECONDARY OUTCOMES:
C-reactive Protein and IL-6 | baseline
fasting blood glucose, lipid profiles | baseline
C-reactive Protein and IL-6 | 6 weeks
fasting blood glucose, lipid profiles | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Po See Chen, MD, Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- National Cheng-Kung University Hospital, Tainan, Taiwan